CLINICAL TRIAL: NCT06792552
Title: A Phase I First-in-human, Open-label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0505 in Adult Participants With Advanced Solid Tumors
Brief Title: A Phase I Study of SIM0505 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NextCure, Inc. (Industry)
Collaborators: Shanghai Xianxiang Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0505-101
Record Dates: First submitted 2025-01-13; First posted 2025-01-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SIM0505 mono dose escalation (Experimental): Every 21 days is one cycle. Multiple dose levels of SIM0505 will be explored in dose escalation, and determine the maximum tolerated dose.
  Interventions: Drug: SIM0505 for injection
- SIM0505 mono dose optimization - Ovarian (Experimental): Every 21 days is one cycle. 2-3 dose levels of SIM0505 will be explored in dose optimization, and determine the recommended dose (RD) of SIM0505 and evaluate the preliminary anti-tumor activity of SIM0505 in ovarian cancer.
  Interventions: Drug: SIM0505 for injection
- SIM0505 mono dose optimization - Renal (Experimental): Every 21 days is one cycle. 2 dose levels of SIM0505 will be explored in dose optimization, and determine the recommended dose (RD) of SIM0505 and evaluate the preliminary anti-tumor activity of SIM0505 in renal cancer.
  Interventions: Drug: SIM0505 for injection
- SIM0505 mono dose optimization - USC (Experimental): Every 21 days is one cycle. 2 dose levels of SIM0505 will be explored in dose optimization, and determine the recommended dose (RD) of SIM0505 and evaluate the preliminary anti-tumor activity of SIM0505 in uterine cancer.
  Interventions: Drug: SIM0505 for injection
- SIM0505 mono dose optimization - NSCLC (Experimental): Every 21 days is one cycle. 2 dose levels of SIM0505 will be explored in dose optimization, and determine the recommended dose (RD) of SIM0505 and evaluate the preliminary anti-tumor activity of SIM0505 in lung cancer.
  Interventions: Drug: SIM0505 for injection

INTERVENTIONS:
Drug: SIM0505 for injection — Every 21 days is one cycle. Multiple dose levels of SIM0505 will be explored in dose escalation, and determine the maximum tolerated dose.
  Arms: SIM0505 mono dose escalation
Drug: SIM0505 for injection — Every 21 days is one cycle. 2-3 dose levels of SIM0505 will be explored in dose optimization, and determine the recommended dose (RD) of SIM0505 and evaluate the preliminary anti-tumor activity of SIM0505
  Arms: SIM0505 mono dose optimization - NSCLC; SIM0505 mono dose optimization - Ovarian; SIM0505 mono dose optimization - Renal; SIM0505 mono dose optimization - USC

SUMMARY:
This is an open-label, multicenter phase 1 study to evaluate the safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0505 in Adult Participants with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is obtained prior to any procedures that are not considered standard of care
2. ≥18 years of age.
3. In Part 1:

   1. Participants with histologically or cytologically confirmed advanced solid tumors, who have failed or are ineligible for standard of care therapies.
   2. Have progressed on at least one prior systematic anti-tumor regimen, and presence of at least one evaluable lesion according to RECIST Version 1.1. Measurable lesions are required in the backfill period.
   3. In the backfill period, eligible tumor types are limited to high-grade serous ovarian cancer, high-grade endometrioid ovarian cancer, USC, clear cell RCC, papillary RCC and adenocarcinoma of NSCLC without actionable mutation of epidermal growth factor receptor (EGFR). For participants with NSCLC, presence of CDH6 expression through immunohistochemical examination of tumor tissue by central laboratory is required.
4. In Part 2: Participants must have a diagnosis of specific type of metastatic or locally advanced solid tumors and have progressed on or cannot benefit from the most recent systematic anti-tumor regimen (unless otherwise specified), with presence of at least one measurable lesion according to RECIST Version 1.1.

Platinum-resistant ovarian cancer cohort:

a. Participants with histologically or cytologically confirmed high-grade serous ovarian cancer, high-grade endometrioid ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.

Renal cell carcinoma cohort:

a. Participants with histologically- or cytologically-confirmed clear cell RCC or papillary RCC.

Uterine serous carcinoma cohort:

a. Participants with histologically- or cytologically-confirmed USC.

Non-Small Cell Lung Cancer cohort:

1. Participants with histologically- or cytologically-confirmed adenocarcinoma of NSCLC without actionable mutation of EGFR.
2. Presence of CDH6 expression through immunohistochemical examination of tumor tissue.

   5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

   6. Life expectancy of ≥12 weeks. 7. Have adequate organ function as indicated by the laboratory values listed within the protocol.

   8. Women of childbearing potential (WOCBP)must have a negative serum pregnancy test within 72 hours prior to the start of study treatment. WOCBP or male participants are required to use highly effective contraceptive methods , and agree to refrain from donating sperm/egg from signing of informed consent through 180 days after the last dose of study treatment.

   9. Able to provide tumor tissue sample (archival or newly obtained core or excisional biopsy) at biomarker-screening (for NSCLC in both Part 1 and 2) or screening (for non-NSCLC in Part 1) visit of a tumor lesion not previously irradiated for CDH6 testing.

   Exclusion Criteria:
   1. For Part 2: has clear cell, mucinous or sarcomatous histology, mixed tumors containing any histology, or low-grade/borderline ovarian cancer; mixed nonsmall cell and small cell carcinoma, or adenosquamous cell lung cancer with an adenocarcinoma component <50% (the participant is eligible if the adenocarcinoma component is ≥50%).
   2. Any other malignancy within 2 years prior to the first dose of the study treatment except for localized cancers that are considered to have been cured and in the opinion of the Investigator present a low risk for recurrence.
   3. Participant has symptomatic central nervous system (CNS) metastases, or CNS metastases requiring CNS-directed local therapy (such as radiotherapy or surgery) or corticosteroids therapy within 2 weeks of first dose of study treatment.
   4. History of bowel obstruction within 3 months prior to the first dose of study treatment.
   5. Known psychiatric disorder or drug abuse that would interfere the study requirements.
   6. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring drainage or medical intervention within 4 weeks before the first dose of study treatment.
   7. Any active infection requires systemic treatment via intravenous infusion within 2 weeks prior to the first dose of study treatment.
   8. History of non-infectious pneumonitis that has required a course of oral or intravenous steroids to assist with recovery, or interstitial lung disease (ILD) or severe obstructive pulmonary disease.
   9. Prior exposure to other CDH6-targeted agents or an ADC with a topoisomerase I inhibitor payload (e.g., raludotatug deruxtecan/DS-6000).

   12. Major surgery within 2 weeks of receiving the first dose of study treatment.

   13. Has received prior anti-cancer therapies within the following time frames prior to the first dose of study treatment; Previous cytotoxic therapy, anticancer targeted small molecules (e.g., tyrosine kinase inhibitors), hormonal agents within 2 weeks, Anti-cancer antibody or ADC within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of study treatment, Chinese medicines/herbal preparations with anticancer indication taken within 2 weeks and/or Radiation therapy <4 weeks.

   14. Use of any live vaccine therapy within 4 weeks prior to the first dose of study treatment.

   15. Administration of below medications≤14 days prior to the first dose of SIM0505; Strong and moderate CYP3A4 inhibitors and Drugs with known risk of Torsades de Pointes (TdP).

   16. Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS).

   17. Active hepatitis B or hepatitis C infection 18. Participants with clinically significant cardiovascular diseases. 19. History of allogeneic organ transplantation or graft-versus-host disease. 20. Known hypersensitivity to study drug or any of the excipients. 21. Participant is pregnant or breastfeeding. 22. Other conditions that researchers consider inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
dose escalation: Dose-limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 21 days)
dose escalation: Adverse events (AEs) | the whole dose escalation phase，an average of 2 year
dose optimization：Objective response rate (ORR) | the whole dose optimization phase，an average of 1.5 year

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - Sarah Cannon Research Institute (SCRI) - Lake Nona, Orlando, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - University Medical Center of New Orleans LSU-LCMC Health Cancer Center, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Sarah Cannon Research Institute (SCRI) - Nashville, Nashville, Tennessee
  - UT Health San Antonio - Mays Cancer Center, San Antonio, Texas
- China (8):
  - The first medical center of PLA general hospital, Beijing, Beijing Municipality
  - Liaoning Cancer Hospital & Institute, Shenyang, China
  - The Fourth Hospital of Hebei Medical University (Heibei Tumor Hospital), Shijiazhuang, China
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - HunanCancer Hospital, Changsha, Hunan
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No